CLINICAL TRIAL: NCT00200603
Title: Autograft Versus Calcium Phosphate Macroporous Bioceramics as Bone Substitute for Tibial Valgus Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/99/3-G
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2004-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: Calcium phosphate ceramic; tibial osteotomy; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

INTERVENTIONS:
Device: calcium phosphate macroporous bioceramics

SUMMARY:
The aim of the study is to compare radiological behavior of blocks of macroporous phosphocalcium as bone substitute in comparison with iliac crest autograft in tibial valgus osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis eligible for tibial valgus osteotomy
* > 18 y.o

Exclusion Criteria:

* prior tibial osteotomy
* history of local infection
* rheumatoid and other inflammatory arthritis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1999-05

PRIMARY OUTCOMES:
Radiological healing and stability of the osteotomy measure at 3, 6, 12 and 24 months after surgery

SECONDARY OUTCOMES:
Knee and iliac crest painSurgical complicationsFonctional results

CONTACTS AND LOCATIONS:
Overall Officials: François Gouin, MD, Principal Investigator — Nantes UH
Locations (1):
- Gouin François, Nantes, France